CLINICAL TRIAL: NCT05936658
Title: A Multi-center, Open-label, Single Arm Phase III Clinical Trial for the Diagnostic Efficacy Assessment and Safety Evaluation by [18F]Florastamin PET/CT Imaging Examination in Patients With Suspected Recurrent or Metastatic Prostate Cancer
Brief Title: [18F]Florastamin PET/CT Imaging Examination in Patients With Suspected Recurrent or Metastatic Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: FutureChem (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FC303-3-2
Record Dates: First submitted 2023-06-21; First posted 2023-07-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: High Risk Prostate Carcinoma
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The positive predictive values (PPV) of [18F]Florastamin PET/CT imaging (Other): The positive predictive values (PPV) of [18F]Florastamin PET/CT imaging for the detection of recurrent or metastatic prostate cancer in subjects are evaluated.
  Interventions: Drug: [F-18]Florastamin

INTERVENTIONS:
Drug: [F-18]Florastamin — A single dose of [F-18]Florastamin at 10 ± 1 mCi is intravenously administered only to the subjects who meet the inclusion/exclusion criteria, and then [F-18]Florastamin PET/CT imaging is performed from the head to thigh after 105 ± 15 minutes (care should be taken to prevent extravasation of the radiopharmaceutical product).

SUMMARY:
This is a multi-center, open-label, single arm Phase III clinical trial for the diagnostic efficacy assessment and safety evaluation by [18F]Florastamin PET/CT imaging examination to determine the presence of recurrent or metastatic prostate cancer in patients whose recurrent or metastatic lesions have been confirmed through the conventional imaging.

DETAILED DESCRIPTION:
In this study, the diagnostic efficacy of [18F]Florastamin PET/CT imaging at detecting recurrent or metastatic prostate cancer will be evaluated according to the histopathology truth standard in prostate cancer patients whose recurrent or metastatic lesions have been confirmed with the conventional imaging.

Patients who meet the inclusion/exclusion criteria of the clinical study protocol will be enrolled, who then will undergo a biopsy or pelvic lymph node dissection (PLND) for one or more lesion locations confirmed with the conventional imaging within 28 days from [18F]Florastamin PET/CT scanning. After the biopsy or PLND, follow-up will be carried out for 2 weeks. However, if necessary, based on the judgment of the principal investigator, additional visits may be made.

1. Baseline Procedures At the baseline visit, the conventional imaging will be performed. The results of whole-body bone scan and gadolinium-enhanced MRI (for the chest, abdomen or pelvis) within 6 weeks prior to [18F]Florastamin PET/CT scanning will be collected. All conventional imaging examinations will be evaluated by the study site.

   At the time of whole-body bone scanning, examinations will be performed 2 hours after the contrast agent 99mTc-HDP 20 to 30 mCi is administered intravenously.

   At the time of gadolinium-enhanced MRI scanning (for the chest, abdomen or pelvis), the gadolinium contrast agent (Gadobrix 1 cc/kg) will be administered intravenously.
2. Biopsy and PLND Images collected through the conventional imaging during the baseline visit can be selectively used for images to guide a biopsy, and images to decide on biopsy sites will be read by the study site. If more than one legions are identified through the image reading, an intermediary radiology specialist will choose a lesion for which to perform a biopsy; however, among the lesions identified, the one determined to be safe for the subject in the investigator's judgment will be preferred as a site on which to perform a biopsy or PLND, and the final biopsy site will be decided after checking its justification through consultation with the intermediary Department of Radiology.

   A biopsy can be performed while hospitalized, if necessary. Pelvic lymph node dissection (PLND) is surgery to remove the lymph nodes from the pelvis, which is part of a radical prostatectomy, so it is typically performed with hospitalization.
3. Florastamin PET imaging (PSMA-PET Imaging) Uptake values of [18F]Florastamin in the region of interest (ROI) of Florastamin PET imaging are evaluated by an independent evaluator. The independent evaluator records all uptake values observed in the lesion, and analyzes uptake values in the lesion where the biopsy has been performed during analysis of efficacy evaluation.
4. Biopsy and Histopathology Tissues removed through a biopsy or PLND are delivered to the Department of Pathology in accordance with the guidelines of the study site and slides by biopsy or PLND site are produced. A pathologist at the study site performs histopathological evaluation of the slides produced with blinded to results of [18F]Florastamin PET/CT examinations. An area on which a biopsy or PLND has been performed and histopathological results thereof are collected in the eCRF.
5. Histopathology truth standard Tissues removed with a standard method in more than one lesion locations confirmed by the conventional imaging performed prior to [18F]Florastamin PET/CT scanning are evaluated in terms of whether there is prostate cancer, there are any other tumors, it is impossible to read, etc. In addition, the positive/negative result of [18F]Florastamin PET/CT imaging in the applicable location is evaluated by an independent evaluator.

ELIGIBILITY:
Inclusion Criteria:

1. Male aged 19 and older
2. Patients histopathologically diagnosed with prostate cancer
3. Patients who can undergo a percutaneous biopsy or PLND for more than one lesion locations with locally recurrent, new or advanced metastasis as confirmed by MRI or whole-body bone scan performed within 6 weeks prior to screening
4. Patients whose survival is expected to be at least 6 months with ECOG Performance Status ≤ 2
5. Those whose ICF was signed by themselves or their legal guardian or representative after sufficient explanation was given by the investigator about the study objectives, details, characteristics of the investigational device, etc. before enrolled for the study.

Exclusion Criteria:

1. Subjects who have the following disease within 6 months prior to screening:

   * Heart failure that falls into Class III or IV heart failure classified by New York Heart Association;
   * Embolism pulmonary, acute coronary syndrome (unstable angina or myocardial infarction);
   * Acute severe respiratory syndrome;
   * Cerebrovascular disease such as stroke;
   * Uncontrollable hypertension (SBP > 160 mmHg or DBP > 90 mmHg);
   * Uncontrollable heart arrhythmia;
   * Blood clotting disorder.
2. Patients who are receiving radiation therapy or ablative therapy on the prostate bed within 12 weeks prior to screening
3. Patients whose method of systemic treatment for prostate cancer (e.g., hormone therapy, biological therapy, radiation therapy, or chemotherapy) has changed within 3 months prior to screening, or who have to change orstart systemic treatment for prostate cancer while the study is being conducted (until before a biopsy or PLND) However, when systemic treatment has changed into watchful waiting, the patient can participate in the study.
4. According to the laboratory test results, patients who meet the following criteria:

   * Platelet counts (PLT) < 50,000/μL;
   * Serum creatinine > 1.8 mg/dL or eGFR (or GFR) < 30 mL/min/1.7 m2;
   * AST and ALT > 2.5 x upper limit of normal (ULN) (however, for a patient whose hepatic metastasis has been confirmed, AST and ALT > 5 x ULN).
5. Subjects who are suffering from active infectious disease at screening and determined unfit to participate in this study;
6. Subjects with solid tumors other than prostate cancer or hematologic malignancies including lymphoma within 3 years prior to screening (however, they can be enrolled in the case of properly treated non-melanoma skin cancer)
7. Subjects who received gamma-emitting radioactive isotopes of high energy (> 300 keV) within the period 5 times longer than the half-life of this investigational product (about 10 hours) prior to screening
8. Subjects with hypersensitivity to radioisotopes
9. Subjects who participate in other clinical studies that may affect image obtainment from [18F]Florastamin-PET/CT or safety evaluation following IV injection of [18F]Florastamin from the time of enrollment for this study until the end (however, they can be enrolled if participating in a cohort clinical study conducted mainly through simple follow-up without administration of IP from the time of enrollment for the study until the end)
10. Subjects who cannot undergo necessary imaging examinations due to medical conditions or other conditions (serious claustrophobia, radiophobia, etc.) that undermine the subject safety or compliance status for generating reliable data or completing the study in the principal investigator's judgment

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male aged 19 and older
Enrollment: 138 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The positive predictive values(PPV) Evaluation of [18F]Florastamine PET/CT | [18F]Florastamin PET/CT conducts at V2(1 Day/Efficacy & Safety evaluation). Biopy or PLND conducts V3(1Day ~ 28Day/Efficacy & Safety evaluation).
  The positive predictive values (PPV) of [18F]Florastamin PET/CT imaging for the detection of recurrent or metastatic prostate cancer in subjects are evaluated. The PPV is calculated by TP/(TP+FP) x 100% for patients with positive [ 18F]Florastamin PET/CT. True positive is defined as being determined to be positive for prostate cancer according to histopathological results of tissues removed from [18F]Florastamin PET/CT and a biopsy or PLND. False positive is defined as being determined negative for prostate cancer according to the histopathological results of tissues removed through a biopsy or PLND, but determined positive for prostate cancer by [18F]Florastamin PET/CT.

SECONDARY OUTCOMES:
Detection rates of [18F]Florastamin PET/CT imaging | [18F]Florastamin PET/CT conducts at V2(1 Day/Efficacy & Safety evaluation). Biopy or PLND conducts V3(1Day ~ 28Day/Efficacy & Safety evaluation).
  Detection rates of [18F]Florastamin PET/CT imaging in the lesion location (prostate, bones, lymph nodes (inside and outside the pelvis), soft tissues, etc.) are evaluated. Detection rates of [18F]Florastamin PET/CT imaging are defined as the percentage of subjects who have tested positive according to the [18F]Florastamin PET/CT imaging results in any random lesion location such as prostate, bones, lymph nodes (inside and outside the pelvis), and soft tissues.
The sensitivity of [18F]Florastamin PET/CT imaging | [18F]Florastamin PET/CT conducts at V2(1 Day/Efficacy & Safety evaluation). Biopy or PLND conducts V3(1Day ~ 28Day/Efficacy & Safety evaluation).
  The sensitivity of [18F]Florastamin PET/CT imaging for the detection of recurrent or metastatic prostate cancer in subjects is evaluated. The sensitivity is calculated by TP/(TP+FN) x 100% for patients with positive [18F]Florastamin PET/CT. True positive is defined as being determined to be positive for prostate cancer according to [ 18F]Florastamin PET/CT and histopathological results. False positive is defined as being determined negative for prostate cancer according to the histopathological results but determined positive for prostate cancer by [18F]Florastamin PET/CT.
The positive predictive values (PPV) Comparison of [18F]Florastamin PET/CT imaging and conventional imaging | [18F]Florastamin PET/CT conducts at V2(1 Day/Efficacy & Safety evaluation). Biopy or PLND conducts V3(1Day ~ 28Day/Efficacy & Safety evaluation).
  The positive predictive values (PPV) of [18F]Florastamin PET/CT imaging and of the conventional imaging (whole-body bone scan, CT, MRI or ultrasound) are compared and evaluated to detect recurrent or metastatic prostate cancer in subjects.
Evaluation of the standard uptake values of [18F]Florastamin in the lesion location | [18F]Florastamin PET/CT conducts at V2(1 Day/Efficacy & Safety evaluation). Biopy or PLND conducts V3(1Day ~ 28Day/Efficacy & Safety evaluation).
  Standard uptake values (SUVpeak, SUVmax, and SUVr) of [18F]Florastamin for each lesion location (prostate, bones, lymph nodes (inside and outside the pelvis), soft tissues, etc.) decided on by the independent evaluator according to the histopathological results (positive and negative for prostate cancer) are evaluated.
Percentage of subjects who found a different lesion in conventional imaging | Conventional imaging conduct at V1(-42 Days ~ 1 Days). [18F]Florastamin PET/CT conducts at V2(1 Day/Efficacy & Safety evaluation). Biopy or PLND conducts V3(1Day ~ 28Day/Efficacy & Safety evaluation).
  The percentage of subjects who have a different lesion location found by [18F]Florastamin PET/CT that was not identified through the conventional imaging but a biopsy conducted there has confirmed the lesion is evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Young Joung, Ph.D, Principal Investigator — National Cancer Center
Locations (6):
- South Korea (6):
  - National Cancer Center, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ewha womans university mokdong medical center, Soeul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amling CL, Blute ML, Bergstralh EJ, Seay TM, Slezak J, Zincke H. Long-term hazard of progression after radical prostatectomy for clinically localized prostate cancer: continued risk of biochemical failure after 5 years. J Urol. 2000 Jul;164(1):101-5. PMID 10840432
- [Background] Antonarakis ES, Feng Z, Trock BJ, Humphreys EB, Carducci MA, Partin AW, Walsh PC, Eisenberger MA. The natural history of metastatic progression in men with prostate-specific antigen recurrence after radical prostatectomy: long-term follow-up. BJU Int. 2012 Jan;109(1):32-9. doi: 10.1111/j.1464-410X.2011.10422.x. Epub 2011 Jul 20. PMID 21777360
- [Background] Bach-Gansmo T, Nanni C, Nieh PT, Zanoni L, Bogsrud TV, Sletten H, Korsan KA, Kieboom J, Tade FI, Odewole O, Chau A, Ward P, Goodman MM, Fanti S, Schuster DM, Willoch F. Multisite Experience of the Safety, Detection Rate and Diagnostic Performance of Fluciclovine (18F) Positron Emission Tomography/Computerized Tomography Imaging in the Staging of Biochemically Recurrent Prostate Cancer. J Urol. 2017 Mar;197(3 Pt 1):676-683. doi: 10.1016/j.juro.2016.09.117. Epub 2016 Oct 13. PMID 27746282
- [Background] Bauman G, Martin P, Thiessen JD, Taylor R, Moussa M, Gaed M, Rachinsky I, Kassam Z, Chin J, Pautler S, Lee TY, Valliant JF, Ward A. [18F]-DCFPyL Positron Emission Tomography/Magnetic Resonance Imaging for Localization of Dominant Intraprostatic Foci: First Experience. Eur Urol Focus. 2018 Sep;4(5):702-706. doi: 10.1016/j.euf.2016.10.002. Epub 2016 Oct 26. PMID 28753797
- [Background] Blomqvist L, Carlsson S, Gjertsson P, Heintz E, Hultcrantz M, Mejare I, Andren O. Limited evidence for the use of imaging to detect prostate cancer: a systematic review. Eur J Radiol. 2014 Sep;83(9):1601-6. doi: 10.1016/j.ejrad.2014.06.028. Epub 2014 Jul 5. PMID 25059597
- [Background] Bluemel C, Krebs M, Polat B, Linke F, Eiber M, Samnick S, Lapa C, Lassmann M, Riedmiller H, Czernin J, Rubello D, Bley T, Kropf S, Wester HJ, Buck AK, Herrmann K. 68Ga-PSMA-PET/CT in Patients With Biochemical Prostate Cancer Recurrence and Negative 18F-Choline-PET/CT. Clin Nucl Med. 2016 Jul;41(7):515-21. doi: 10.1097/RLU.0000000000001197. PMID 26975008
- [Background] Calais J, Ceci F, Eiber M, Hope TA, Hofman MS, Rischpler C, Bach-Gansmo T, Nanni C, Savir-Baruch B, Elashoff D, Grogan T, Dahlbom M, Slavik R, Gartmann J, Nguyen K, Lok V, Jadvar H, Kishan AU, Rettig MB, Reiter RE, Fendler WP, Czernin J. 18F-fluciclovine PET-CT and 68Ga-PSMA-11 PET-CT in patients with early biochemical recurrence after prostatectomy: a prospective, single-centre, single-arm, comparative imaging trial. Lancet Oncol. 2019 Sep;20(9):1286-1294. doi: 10.1016/S1470-2045(19)30415-2. Epub 2019 Jul 30. PMID 31375469
- [Background] Calais J, Fendler WP, Herrmann K, Eiber M, Ceci F. Comparison of 68Ga-PSMA-11 and 18F-Fluciclovine PET/CT in a Case Series of 10 Patients with Prostate Cancer Recurrence. J Nucl Med. 2018 May;59(5):789-794. doi: 10.2967/jnumed.117.203257. Epub 2017 Dec 14. PMID 29242404
- [Background] Castellucci P, Fuccio C, Nanni C, Santi I, Rizzello A, Lodi F, Franceschelli A, Martorana G, Manferrari F, Fanti S. Influence of trigger PSA and PSA kinetics on 11C-Choline PET/CT detection rate in patients with biochemical relapse after radical prostatectomy. J Nucl Med. 2009 Sep;50(9):1394-400. doi: 10.2967/jnumed.108.061507. Epub 2009 Aug 18. PMID 19690023
- [Background] Chang SS. Overview of prostate-specific membrane antigen. Rev Urol. 2004;6 Suppl 10(Suppl 10):S13-8. PMID 16985927
- [Background] Chausse G, Niazi T, Abikhzer GS, Probst SM. Biopsy-Proven Diffuse Mediastinal Prostate Cancer Metastases Negative on 18F-Fluorocholine, Diagnosed on 68Ga-PSMA and 18F-PSMA PET/CT. Clin Nucl Med. 2017 Oct;42(10):801-802. doi: 10.1097/RLU.0000000000001766. PMID 28719448
- [Background] Chen Y, Pullambhatla M, Foss CA, Byun Y, Nimmagadda S, Senthamizhchelvan S, Sgouros G, Mease RC, Pomper MG. 2-(3-1-Carboxy-5-[(6-[18F]fluoro-pyridine-3-carbonyl)-amino]-pentyl-ureido)-pentanedioic acid, [18F]DCFPyL, a PSMA-based PET imaging agent for prostate cancer. Clin Cancer Res. 2011 Dec 15;17(24):7645-53. doi: 10.1158/1078-0432.CCR-11-1357. Epub 2011 Oct 31. PMID 22042970
- [Background] de Jong IJ, Pruim J, Elsinga PH, Vaalburg W, Mensink HJ. 11C-choline positron emission tomography for the evaluation after treatment of localized prostate cancer. Eur Urol. 2003 Jul;44(1):32-8; discussion 38-9. doi: 10.1016/s0302-2838(03)00207-0. PMID 12814672
- [Background] Dietlein M, Kobe C, Kuhnert G, Stockter S, Fischer T, Schomacker K, Schmidt M, Dietlein F, Zlatopolskiy BD, Krapf P, Richarz R, Neubauer S, Drzezga A, Neumaier B. Comparison of [(18)F]DCFPyL and [ (68)Ga]Ga-PSMA-HBED-CC for PSMA-PET Imaging in Patients with Relapsed Prostate Cancer. Mol Imaging Biol. 2015 Aug;17(4):575-84. doi: 10.1007/s11307-015-0866-0. PMID 26013479
- [Background] Eiber M, Maurer T, Souvatzoglou M, Beer AJ, Ruffani A, Haller B, Graner FP, Kubler H, Haberkorn U, Eisenhut M, Wester HJ, Gschwend JE, Schwaiger M. Evaluation of Hybrid (6)(8)Ga-PSMA Ligand PET/CT in 248 Patients with Biochemical Recurrence After Radical Prostatectomy. J Nucl Med. 2015 May;56(5):668-74. doi: 10.2967/jnumed.115.154153. Epub 2015 Mar 19. PMID 25791990
- [Background] Evangelista L, Briganti A, Fanti S, Joniau S, Reske S, Schiavina R, Stief C, Thalmann GN, Picchio M. New Clinical Indications for (18)F/(11)C-choline, New Tracers for Positron Emission Tomography and a Promising Hybrid Device for Prostate Cancer Staging: A Systematic Review of the Literature. Eur Urol. 2016 Jul;70(1):161-175. doi: 10.1016/j.eururo.2016.01.029. Epub 2016 Feb 2. PMID 26850970
- [Background] Fendler WP, Calais J, Eiber M, Flavell RR, Mishoe A, Feng FY, Nguyen HG, Reiter RE, Rettig MB, Okamoto S, Emmett L, Zacho HD, Ilhan H, Wetter A, Rischpler C, Schoder H, Burger IA, Gartmann J, Smith R, Small EJ, Slavik R, Carroll PR, Herrmann K, Czernin J, Hope TA. Assessment of 68Ga-PSMA-11 PET Accuracy in Localizing Recurrent Prostate Cancer: A Prospective Single-Arm Clinical Trial. JAMA Oncol. 2019 Jun 1;5(6):856-863. doi: 10.1001/jamaoncol.2019.0096. PMID 30920593
- [Background] Ghosh A, Heston WD. Tumor target prostate specific membrane antigen (PSMA) and its regulation in prostate cancer. J Cell Biochem. 2004 Feb 15;91(3):528-39. doi: 10.1002/jcb.10661. PMID 14755683
- [Background] Giovacchini G, Picchio M, Coradeschi E, Scattoni V, Bettinardi V, Cozzarini C, Freschi M, Fazio F, Messa C. [(11)C]choline uptake with PET/CT for the initial diagnosis of prostate cancer: relation to PSA levels, tumour stage and anti-androgenic therapy. Eur J Nucl Med Mol Imaging. 2008 Jun;35(6):1065-73. doi: 10.1007/s00259-008-0716-2. Epub 2008 Jan 16. PMID 18200444
- [Background] Gorin MA, Rowe SP, Patel HD, Vidal I, Mana-Ay M, Javadi MS, Solnes LB, Ross AE, Schaeffer EM, Bivalacqua TJ, Partin AW, Pienta KJ, Szabo Z, De Marzo AM, Pomper MG, Allaf ME. Prostate Specific Membrane Antigen Targeted 18F-DCFPyL Positron Emission Tomography/Computerized Tomography for the Preoperative Staging of High Risk Prostate Cancer: Results of a Prospective, Phase II, Single Center Study. J Urol. 2018 Jan;199(1):126-132. doi: 10.1016/j.juro.2017.07.070. Epub 2017 Jul 20. PMID 28736318
- [Background] Greco C, Cascini GL, Tamburrini O. Is there a role for positron emission tomography imaging in the early evaluation of prostate cancer relapse? Prostate Cancer Prostatic Dis. 2008;11(2):121-8. doi: 10.1038/sj.pcan.4501028. Epub 2008 Jan 8. PMID 18180806
- [Background] Han M, Partin AW, Zahurak M, Piantadosi S, Epstein JI, Walsh PC. Biochemical (prostate specific antigen) recurrence probability following radical prostatectomy for clinically localized prostate cancer. J Urol. 2003 Feb;169(2):517-23. doi: 10.1097/01.ju.0000045749.90353.c7. PMID 12544300
- [Background] Hillier SM, Maresca KP, Femia FJ, Marquis JC, Foss CA, Nguyen N, Zimmerman CN, Barrett JA, Eckelman WC, Pomper MG, Joyal JL, Babich JW. Preclinical evaluation of novel glutamate-urea-lysine analogues that target prostate-specific membrane antigen as molecular imaging pharmaceuticals for prostate cancer. Cancer Res. 2009 Sep 1;69(17):6932-40. doi: 10.1158/0008-5472.CAN-09-1682. Epub 2009 Aug 25. PMID 19706750
- [Background] Hillier SM, Maresca KP, Lu G, Merkin RD, Marquis JC, Zimmerman CN, Eckelman WC, Joyal JL, Babich JW. 99mTc-labeled small-molecule inhibitors of prostate-specific membrane antigen for molecular imaging of prostate cancer. J Nucl Med. 2013 Aug;54(8):1369-76. doi: 10.2967/jnumed.112.116624. Epub 2013 Jun 3. PMID 23733925
- [Background] Hofer C, Laubenbacher C, Block T, Breul J, Hartung R, Schwaiger M. Fluorine-18-fluorodeoxyglucose positron emission tomography is useless for the detection of local recurrence after radical prostatectomy. Eur Urol. 1999;36(1):31-5. doi: 10.1159/000019923. PMID 10364652
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Kinoshita Y, Kuratsukuri K, Landas S, Imaida K, Rovito PM Jr, Wang CY, Haas GP. Expression of prostate-specific membrane antigen in normal and malignant human tissues. World J Surg. 2006 Apr;30(4):628-36. doi: 10.1007/s00268-005-0544-5. PMID 16555021
- [Background] Krause BJ, Souvatzoglou M, Tuncel M, Herrmann K, Buck AK, Praus C, Schuster T, Geinitz H, Treiber U, Schwaiger M. The detection rate of [11C]choline-PET/CT depends on the serum PSA-value in patients with biochemical recurrence of prostate cancer. Eur J Nucl Med Mol Imaging. 2008 Jan;35(1):18-23. doi: 10.1007/s00259-007-0581-4. Epub 2007 Sep 22. PMID 17891394
- [Background] Li X, Rowe SP, Leal JP, Gorin MA, Allaf ME, Ross AE, Pienta KJ, Lodge MA, Pomper MG. Semiquantitative Parameters in PSMA-Targeted PET Imaging with 18F-DCFPyL: Variability in Normal-Organ Uptake. J Nucl Med. 2017 Jun;58(6):942-946. doi: 10.2967/jnumed.116.179739. Epub 2016 Dec 8. PMID 27932557
- [Background] Mena E, Lindenberg ML, Turkbey IB, Shih JH, Harmon SA, Lim I, Lin F, Adler S, Eclarinal P, McKinney YL, Citrin D, Dahut W, Wood BJ, Krishnasamy V, Chang R, Levy E, Merino M, Pinto P, Eary JF, Choyke PL. 18F-DCFPyL PET/CT Imaging in Patients with Biochemically Recurrent Prostate Cancer After Primary Local Therapy. J Nucl Med. 2020 Jun;61(6):881-889. doi: 10.2967/jnumed.119.234799. Epub 2019 Nov 1. PMID 31676732
- [Background] Morris MJ, Rowe SP, Gorin MA, Saperstein L, Pouliot F, Josephson D, Wong JYC, Pantel AR, Cho SY, Gage KL, Piert M, Iagaru A, Pollard JH, Wong V, Jensen J, Lin T, Stambler N, Carroll PR, Siegel BA; CONDOR Study Group. Diagnostic Performance of 18F-DCFPyL-PET/CT in Men with Biochemically Recurrent Prostate Cancer: Results from the CONDOR Phase III, Multicenter Study. Clin Cancer Res. 2021 Jul 1;27(13):3674-3682. doi: 10.1158/1078-0432.CCR-20-4573. Epub 2021 Feb 23. PMID 33622706
- [Background] Nanni C, Zanoni L, Pultrone C, Schiavina R, Brunocilla E, Lodi F, Malizia C, Ferrari M, Rigatti P, Fonti C, Martorana G, Fanti S. (18)F-FACBC (anti1-amino-3-(18)F-fluorocyclobutane-1-carboxylic acid) versus (11)C-choline PET/CT in prostate cancer relapse: results of a prospective trial. Eur J Nucl Med Mol Imaging. 2016 Aug;43(9):1601-10. doi: 10.1007/s00259-016-3329-1. Epub 2016 Mar 10. PMID 26960562
- [Background] Nunez R, Macapinlac HA, Yeung HW, Akhurst T, Cai S, Osman I, Gonen M, Riedel E, Scher HI, Larson SM. Combined 18F-FDG and 11C-methionine PET scans in patients with newly progressive metastatic prostate cancer. J Nucl Med. 2002 Jan;43(1):46-55. PMID 11801702
- [Background] Odewole OA, Tade FI, Nieh PT, Savir-Baruch B, Jani AB, Master VA, Rossi PJ, Halkar RK, Osunkoya AO, Akin-Akintayo O, Zhang C, Chen Z, Goodman MM, Schuster DM. Recurrent prostate cancer detection with anti-3-[(18)F]FACBC PET/CT: comparison with CT. Eur J Nucl Med Mol Imaging. 2016 Sep;43(10):1773-83. doi: 10.1007/s00259-016-3383-8. Epub 2016 Apr 18. PMID 27091135
- [Background] Perner S, Hofer MD, Kim R, Shah RB, Li H, Moller P, Hautmann RE, Gschwend JE, Kuefer R, Rubin MA. Prostate-specific membrane antigen expression as a predictor of prostate cancer progression. Hum Pathol. 2007 May;38(5):696-701. doi: 10.1016/j.humpath.2006.11.012. Epub 2007 Feb 22. PMID 17320151
- [Background] Petrylak DP, Tangen CM, Hussain MH, Lara PN Jr, Jones JA, Taplin ME, Burch PA, Berry D, Moinpour C, Kohli M, Benson MC, Small EJ, Raghavan D, Crawford ED. Docetaxel and estramustine compared with mitoxantrone and prednisone for advanced refractory prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1513-20. doi: 10.1056/NEJMoa041318. PMID 15470214
- [Background] Pfister D, Porres D, Heidenreich A, Heidegger I, Knuechel R, Steib F, Behrendt FF, Verburg FA. Detection of recurrent prostate cancer lesions before salvage lymphadenectomy is more accurate with (68)Ga-PSMA-HBED-CC than with (18)F-Fluoroethylcholine PET/CT. Eur J Nucl Med Mol Imaging. 2016 Jul;43(8):1410-7. doi: 10.1007/s00259-016-3366-9. Epub 2016 Mar 19. PMID 26993315
- [Background] Pienta KJ, Gorin MA, Rowe SP, Carroll PR, Pouliot F, Probst S, Saperstein L, Preston MA, Alva AS, Patnaik A, Durack JC, Stambler N, Lin T, Jensen J, Wong V, Siegel BA, Morris MJ. A Phase 2/3 Prospective Multicenter Study of the Diagnostic Accuracy of Prostate Specific Membrane Antigen PET/CT with 18F-DCFPyL in Prostate Cancer Patients (OSPREY). J Urol. 2021 Jul;206(1):52-61. doi: 10.1097/JU.0000000000001698. Epub 2021 Feb 26. PMID 33634707
- [Background] Pinto JT, Suffoletto BP, Berzin TM, Qiao CH, Lin S, Tong WP, May F, Mukherjee B, Heston WD. Prostate-specific membrane antigen: a novel folate hydrolase in human prostatic carcinoma cells. Clin Cancer Res. 1996 Sep;2(9):1445-51. PMID 9816319
- [Background] Pound CR, Partin AW, Eisenberger MA, Chan DW, Pearson JD, Walsh PC. Natural history of progression after PSA elevation following radical prostatectomy. JAMA. 1999 May 5;281(17):1591-7. doi: 10.1001/jama.281.17.1591. PMID 10235151
- [Background] Pucar D, Sella T, Schoder H. The role of imaging in the detection of prostate cancer local recurrence after radiation therapy and surgery. Curr Opin Urol. 2008 Jan;18(1):87-97. doi: 10.1097/MOU.0b013e3282f13ac3. PMID 18090496
- [Background] Reinfelder J, Kuwert T, Beck M, Sanders JC, Ritt P, Schmidkonz C, Hennig P, Prante O, Uder M, Wullich B, Goebell P. First Experience With SPECT/CT Using a 99mTc-Labeled Inhibitor for Prostate-Specific Membrane Antigen in Patients With Biochemical Recurrence of Prostate Cancer. Clin Nucl Med. 2017 Jan;42(1):26-33. doi: 10.1097/RLU.0000000000001433. PMID 27775936
- [Background] Rinnab L, Mottaghy FM, Blumstein NM, Reske SN, Hautmann RE, Hohl K, Moller P, Wiegel T, Kuefer R, Gschwend JE. Evaluation of [11C]-choline positron-emission/computed tomography in patients with increasing prostate-specific antigen levels after primary treatment for prostate cancer. BJU Int. 2007 Oct;100(4):786-93. doi: 10.1111/j.1464-410X.2007.07083.x. PMID 17822459
- [Background] Rowe SP, Macura KJ, Mena E, Blackford AL, Nadal R, Antonarakis ES, Eisenberger M, Carducci M, Fan H, Dannals RF, Chen Y, Mease RC, Szabo Z, Pomper MG, Cho SY. PSMA-Based [(18)F]DCFPyL PET/CT Is Superior to Conventional Imaging for Lesion Detection in Patients with Metastatic Prostate Cancer. Mol Imaging Biol. 2016 Jun;18(3):411-9. doi: 10.1007/s11307-016-0957-6. PMID 27080322
- [Background] Rowe SP, Pienta KJ, Pomper MG, Gorin MA. PSMA-RADS Version 1.0: A Step Towards Standardizing the Interpretation and Reporting of PSMA-targeted PET Imaging Studies. Eur Urol. 2018 Apr;73(4):485-487. doi: 10.1016/j.eururo.2017.10.027. Epub 2017 Nov 11. PMID 29132714
- [Background] Scattoni V, Picchio M, Suardi N, Messa C, Freschi M, Roscigno M, Da Pozzo L, Bocciardi A, Rigatti P, Fazio F. Detection of lymph-node metastases with integrated [11C]choline PET/CT in patients with PSA failure after radical retropubic prostatectomy: results confirmed by open pelvic-retroperitoneal lymphadenectomy. Eur Urol. 2007 Aug;52(2):423-9. doi: 10.1016/j.eururo.2007.03.032. Epub 2007 Mar 20. PMID 17397992
- [Background] Scheidler J, Hricak H, Vigneron DB, Yu KK, Sokolov DL, Huang LR, Zaloudek CJ, Nelson SJ, Carroll PR, Kurhanewicz J. Prostate cancer: localization with three-dimensional proton MR spectroscopic imaging--clinicopathologic study. Radiology. 1999 Nov;213(2):473-80. doi: 10.1148/radiology.213.2.r99nv23473. PMID 10551229
- [Background] Schuster DM, Nieh PT, Jani AB, Amzat R, Bowman FD, Halkar RK, Master VA, Nye JA, Odewole OA, Osunkoya AO, Savir-Baruch B, Alaei-Taleghani P, Goodman MM. Anti-3-[(18)F]FACBC positron emission tomography-computerized tomography and (111)In-capromab pendetide single photon emission computerized tomography-computerized tomography for recurrent prostate carcinoma: results of a prospective clinical trial. J Urol. 2014 May;191(5):1446-53. doi: 10.1016/j.juro.2013.10.065. Epub 2013 Oct 19. PMID 24144687
- [Background] Schuster DM, Votaw JR, Nieh PT, Yu W, Nye JA, Master V, Bowman FD, Issa MM, Goodman MM. Initial experience with the radiotracer anti-1-amino-3-18F-fluorocyclobutane-1-carboxylic acid with PET/CT in prostate carcinoma. J Nucl Med. 2007 Jan;48(1):56-63. PMID 17204699
- [Background] Shreve PD, Grossman HB, Gross MD, Wahl RL. Metastatic prostate cancer: initial findings of PET with 2-deoxy-2-[F-18]fluoro-D-glucose. Radiology. 1996 Jun;199(3):751-6. doi: 10.1148/radiology.199.3.8638000.
- [Background] Silver DA, Pellicer I, Fair WR, Heston WD, Cordon-Cardo C. Prostate-specific membrane antigen expression in normal and malignant human tissues. Clin Cancer Res. 1997 Jan;3(1):81-5. PMID 9815541
- [Background] Smith-Jones PM, Vallabahajosula S, Goldsmith SJ, Navarro V, Hunter CJ, Bastidas D, Bander NH. In vitro characterization of radiolabeled monoclonal antibodies specific for the extracellular domain of prostate-specific membrane antigen. Cancer Res. 2000 Sep 15;60(18):5237-43. PMID 11016653
- [Background] Tannock IF, de Wit R, Berry WR, Horti J, Pluzanska A, Chi KN, Oudard S, Theodore C, James ND, Turesson I, Rosenthal MA, Eisenberger MA; TAX 327 Investigators. Docetaxel plus prednisone or mitoxantrone plus prednisone for advanced prostate cancer. N Engl J Med. 2004 Oct 7;351(15):1502-12. doi: 10.1056/NEJMoa040720. PMID 15470213
- [Background] Thompson IM, Valicenti RK, Albertsen P, Davis BJ, Goldenberg SL, Hahn C, Klein E, Michalski J, Roach M, Sartor O, Wolf JS Jr, Faraday MM. Adjuvant and salvage radiotherapy after prostatectomy: AUA/ASTRO Guideline. J Urol. 2013 Aug;190(2):441-9. doi: 10.1016/j.juro.2013.05.032. Epub 2013 May 21. PMID 23707439
- [Background] Treglia G, Ceriani L, Sadeghi R, Giovacchini G, Giovanella L. Relationship between prostate-specific antigen kinetics and detection rate of radiolabelled choline PET/CT in restaging prostate cancer patients: a meta-analysis. Clin Chem Lab Med. 2014 May;52(5):725-33. doi: 10.1515/cclm-2013-0675. PMID 24310773
- [Background] Troyer JK, Beckett ML, Wright GL Jr. Detection and characterization of the prostate-specific membrane antigen (PSMA) in tissue extracts and body fluids. Int J Cancer. 1995 Sep 4;62(5):552-8. doi: 10.1002/ijc.2910620511. PMID 7665226
- [Background] Wondergem M, van der Zant FM, Knol RJJ, Lazarenko SV, Pruim J, de Jong IJ. 18F-DCFPyL PET/CT in the Detection of Prostate Cancer at 60 and 120 Minutes: Detection Rate, Image Quality, Activity Kinetics, and Biodistribution. J Nucl Med. 2017 Nov;58(11):1797-1804. doi: 10.2967/jnumed.117.192658. Epub 2017 Apr 27. PMID 28450569